CLINICAL TRIAL: NCT04362111
Title: Early Treatment of Cytokine Storm Syndrome in Covid-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, W Winn Chatham, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Chatham-Cytokine Covid-19
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cytokine Storm; COVID-19
MeSH Terms: conditions — Cytokine Release Syndrome; COVID-19 | interventions — Interleukin 1 Receptor Antagonist Protein; Saline Solution

STUDY DESIGN:
Intervention Model Description: Two parallel treatment arms
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigator, care provider, and participant blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anakinra Group (Experimental): The active treatment group will receive anakinra 100 mg subcutaneously every 6 hours for period of 10 days. For subjects meeting complete response criteria at 5 days, dosing will be decreased to 100 mg twice daily for the remaining 5 days.
  Interventions: Drug: Anakinra
- Control Group (Placebo Comparator): The control group will receive normal saline placebo subcutaneously every 6 hours for period of 10 days. For subjects meeting complete response criteria at 5 days, dosing will be decreased to twice daily for the remaining 5 days.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Anakinra — The active treatment group will receive anakinra 100 mg subcutaneously every 6-12 hours for a period of 10 days
  Other Names: recombinant human IL-ra (rhIL-1ra)
  Arms: Anakinra Group
Drug: Normal saline — The control group will receive normal saline placebo subcutaneously every 6-12 hours for period of 10 days
  Other Names: NS
  Arms: Control Group

SUMMARY:
This proposal addresses the problem of preventing the very high mortality and morbidity associated with the development of Cytokine Storm Syndrome (CSS) associated respiratory failure in Covid-19 infection.

DETAILED DESCRIPTION:
The first aim of this project is to determine whether rapidly assayed early clinical laboratory markers of CSS (eCSS: leucopenia, lymphopenia, and elevated ferritin, d-dimer, LDH, CRP, and AST/ALT) in patients admitted to the hospital with respiratory compromise in the setting of Covid-19 infection can accurately identify patients with CSS as defined by validated CSS case definitions (H-Score, aHLH-2004). Confirmation of eCSS predictive of evolving CSS will identify patients at risk for rapid deterioration of lung function and inform early initiation of treatment for CSS. Genotyping studies will also be performed on patients with confirmed CSS to determine whether perforin pathway mutations commonly present in CSS associated with other disorders are present. The second aim is to determine whether early treatment with rhIL-1Ra (anakinra) in patients admitted to the hospital with markers of CSS improves or prevents deterioration of respiratory dysfunction and prevents the development of respiratory failure requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Molecular (pcRNA) diagnosis of SARS-CoV-2 infection
3. Chest imaging studies consistent with Covid-19 pneumonia
4. Hyperferritinemia (>700 ng/ml)
5. History of fever >38 degrees C
6. Any three of the following:

   1. Elevated d-dimer (> 500 ng/ml)
   2. thrombocytopenia (< 130,000/mm3)
   3. leucopenia (WBC <3500/mm3) or lymphopenia (<1000/mm3)
   4. elevated AST or ALT (> 2X ULN)
   5. elevated LDH (> 2X ULN)
   6. CRP > 100 mg/L

Exclusion Criteria:

1. Participation in other investigational treatment protocols for Covid-19 infection
2. Culture confirmed active bacterial infection requiring antibiotic therapy
3. On mechanical ventilation
4. Previous known hypersensitivity reaction to anakinra
5. Previous known hypersensitivity reaction to E Coli derived proteins
6. Pregnant or breast-feeding females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter W Chatham, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI by e-mail for protocol specifics Submission of results for peer reviewed publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: During study enrollment
Access Criteria: wchatham@uabmc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects for enrollment were identified by pre-screening all patients admitted to the University of Alabama Hospital for treatment of Covid-19 pneumonia from August 1, 2020-January 15, 2021. Patients who were admitted with a new requirement for supplemental oxygen to maintain arterial oxygen saturation >93% but not yet requiring mechanical ventilation and who had admission laboratory studies meeting study inclusion criteria for evidence of inflammation were approached for enrollment.
Pre-assignment Details: Patients who met inclusion/exclusion criteria and who had ongoing or increasing oxygen requirement were consented and enrolled. Once consented and enrolled, all subjects were randomly assigned to the two treatment groups. No participants were excluded after enrollment and randomization. Two subjects withdrew consent within 48 hours of enrollment.
Period: Overall Study
Arm/Group | Anakinra Group | Control Group
Started | 15 | 17 (Two patients randomized to the placebo group withdrew within 48 hours of enrollment/randomization. An additional two subjects were enrolled and assigned to the placebo group to balance the treatment groups with regard to participants completing the study. The investigators were blinded as to which group(s) the two subjects withdrawing consent had been randomized to.)
Completed | 15 | 15
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control Group: The control group will receive normal saline placebo subcutaneously every 6 hours for period of 10 days. For subjects meeting complete repsonse criteria at 5 days, dosing wll be decreased to twice daily for the remaining 5 days.
  Normal saline: The control group will receive normal saline placebo subcutaneously every 6-12 hours for period of 10 days
- Total: Total of all reporting groups
Arm/Group | Anakinra Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (8.2) | 61.8 (12.2) | 63.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Co-morbidities [Count of Participants; unit: Participants]
  Cardiovascular Disease | 4 | 3 | 7
  Diabetes | 5 | 3 | 8
  Hypertension | 11 | 10 | 21
Number of Participants that Smoke [Count of Participants; unit: Participants] | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Subjects Discharged From the Hospital Alive and Without the Need for Mechanical Ventilation.
Description: Percentage of subjects discharged from hospital alive and who did not require intubation and mechanical ventilation
Time Frame: Variable up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 10 | 10

2. Secondary Outcome: Percentage of Subjects With 25% Change (Decrease) in Cytokine Storm Markers at 48-72 Hours After Dosing With Study Agent
Description: 25% change (decrease) in noted baseline elevations of serum ferritin and CRP measured 48-72 hours after following initial dosing of anakinra/placebo.
Time Frame: 48 hours after taking initial dose of anakinra/placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 6 | 8

3. Secondary Outcome: Percentage of Subjects Without Increase in Oxygen Requirement and no Increase in Oxygen Delivery/Respiratory Support Measures After 48 Hours.
Description: Supplemental oxygen requirement to maintain oxygen saturation >90% stable or decreased without escalation of respiratory support measures (addition of CPAP, initiation of mechanical ventilation)
Time Frame: Day 2 (48 hours)-Day 10 (240 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 8 | 9

4. Secondary Outcome: Patients Requiring Minimal Oxygen Support at Day 10
Description: Percentage of participants requiring no more than 2 L/min nasal canula oxygen to maintain oxygen saturation >93% by Day 10
Time Frame: 0-10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 8 | 9

5. Secondary Outcome: Percentage of Subjects With Resolution of Laboratory Markers of Cytokine Storm Syndrome
Description: Normalization or ≥ 75% improvement by Day 10 (120 hours) in each (all) of the following laboratory CSS attributes elevated beyond the normal range at randomization: ferritin, d-dimer, CRP, and LDH.
Time Frame: Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 0 | 7

6. Secondary Outcome: Percentage of Subjects Who Develop Bacterial or Fungal or Non-Covid-19 Viral Infection
Description: Occurence of new bacterial or fungal or viral infection through the time of hospital discharge or Day 28.
Time Frame: Day 0-28
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 1 | 0

7. Secondary Outcome: Absence of Supplemental Oxygen Requirement at Day 10
Description: Percentage of participants able to maintain oxygen saturation >93% on room air by Day 10
Time Frame: 0-10 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra Group | Control Group
Number analyzed (Participants) | 15 | 15
Participants | 4 | 9

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Anakinra Group | Control Group
All-Cause Mortality (participants affected / at risk) | 4/15 | 4/15
Serious Adverse Events (participants affected / at risk) | 9/15 | 7/15
Other Adverse Events (participants affected / at risk) | 14/15 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra Group (N=15) | Control Group (N=15)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (9) — Development of respiratory failure due to diffuse lung inflammation
Arterial ischemia (Vascular disorders) | 4 (4) | 5 (5) — Evidence of ischemic injury to an extremity or internal organ or central nervous system
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra Group (N=15) | Control Group (N=15)
Venous thrombosis (Blood and lymphatic system disorders) | 4 (4) | 3 (3) — Deep venous thrombosis, with or without pulmonary embolism
Acute Renal Failure (Renal and urinary disorders) | 7 (7) | 6 (6) — Development of acute kidney injury with azotemia and decreased urine output
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Total neutrophil count less than 1000/mm3
Anemia (Blood and lymphatic system disorders) | 14 (14) | 13 (13) — Decrease in hemoglobin to less than 8.0 g/dL
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 5 (5) — Decrease in platelets to less than 100,000/mm3
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Evidence of clinically significant GI bleed with documented GI blood loss and associated fall in hemoglobin

LIMITATIONS AND CAVEATS:
1. All subjects received daily dexamethasone to the standard of care management of Covid-19 pneumonia requiring hospitalization.
2. Some of the enrolled subjects with rapid improvement were discharged prior to 10 days with instructions on anakinra self-administration at home; adherence with unsupervised dosing of study agent could not be readily assessed, nor could reported oxygen saturations be confirmed in these participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04362111/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04362111/ICF_001.pdf